CLINICAL TRIAL: NCT02505529
Title: Neural Mechanisms of Dynapenia
Brief Title: The UNCODE Study: Unravelling the Neural Contributors Of Dynapenia in Elders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio University (Other)
Collaborators: National Institute on Aging (NIA) (NIH); University of Florida (Other); Holzer Health System (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 14F038; R01AG044424 (NIH)
Record Dates: First submitted 2015-07-20; First posted 2015-07-22 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Aging
Keywords: Aging; Muscle; Weakness; Sarcopenia; Dynapenia
MeSH Terms: conditions — Asthenia; Sarcopenia | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Resistance Exercise Training (Experimental): 12-weeks of high-intensity, progressive resistance exercise training (3x/wk).
  Interventions: Other: Resistance Exercise Training
- Mental Imagery (Experimental): 6-weeks of mental imagery of strong muscle contractions and mobility tasks (5x/wk).
  Interventions: Other: Mental Imagery
- Control Group (No Intervention): 6-weeks of no change in lifestyle.

INTERVENTIONS:
Other: Resistance Exercise Training — Behavioral interventions of resistance exercise
  Arms: Resistance Exercise Training
Other: Mental Imagery — Behavioral intervention of mental imagery
  Arms: Mental Imagery

SUMMARY:
The UNCODE Study seeks to better identify the neurological causes of muscle weakness associated with advancing age. The main study consists of 4 laboratory-based testing sessions that involve testing muscle strength and physical and cognitive function as well as a battery of tests to 1) quantify brain excitability (using non-invasive transcranial magnetic stimulation), 2) modulate brain excitability (using non-invasive transcranial direct current stimulation), 3) spinal motor nerve firing characteristics, and 4) brain structure and function characteristics based on magnetic resonance images of the brain. Additionally, three option sub-studies are also available for enrollment. The first is a genetics sub-study where a cheek swab will be used to examine associations between certain genes and the physiological and functional measures obtained from the main study. The other two sub-studies are interventions. The first sub-study is a progressive resistance exercise training study where study participants will undergo 12-weeks of exercise training (3x/wk) and at the completion of the exercise training the measures obtained in the main study will be re-assessed. The other sub-study is a mental imagery sub-study where subjects are randomly assigned to perform a mental imagery training program consisting of imaging strong muscle contractions and mobility tasks (5x/wk) or to serve as a control (i.e., to not modify lifestyle) for 6-weeks. At the completion of the respective intervention period the measures obtained in the main study will be re-assessed.

DETAILED DESCRIPTION:
The UNCODE Study seeks to better identify the neurological causes of muscle weakness associated with advancing age. The main study consists of 4 laboratory-based testing sessions that involve testing muscle strength and physical and cognitive function as well as a battery of tests to 1) quantify brain excitability (using single and paired pulse transcranial magnetic stimulation of the upper and lower extremity muscles), 2) modulate brain excitability of the upper extremity muscles (using non-invasive transcranial direct current stimulation), 3) spinal motor nerve firing characteristics using decomposition surface electromyography, and 4) brain structure and function characteristics based on magnetic resonance images of the brain. Additionally, three optional sub-studies are also available for enrollment. The first is a genetics sub-study where a cheek swab will be used to examine associations between certain genes (APOE-4 allele) and the physiological and functional measures obtained from the main study. The other two sub-studies are interventions. The first sub-study is a progressive resistance exercise training study where study participants will undergo 12-weeks of exercise training (3x/wk) and at the completion of the exercise training the measures obtained in the main study will be re-assessed. The other sub-study is a mental imagery sub-study where subjects are randomly assigned to perform a mental imagery training program consisting of imaging strong muscle contractions and mobility tasks (5x/wk) or to serve as a control (i.e., to not modify lifestyle) for 6-weeks. At the completion of the respective intervention period the measures obtained in the main study will be re-assessed.

ELIGIBILITY:
Inclusion Criteria:

* Age 60+ years with no significant health issues or conditions that, in the investigator's opinion, would limit the subject's ability to complete the study per protocol or that would impact the capability to get an accurate measurement of study endpoints.
* Body mass index between 16.0 and 40.0 kg/m2.
* With no condition that would limit participation in supervised resistance training exercise based on the Physical Activity Readiness Questionnaire (PAR-Q) (for the "Resistance Exercise Training Sub-Study only).
* Willingness to maintain current diet and adhere to the intervention programs described for the sub-studies (if applicable) and willing to undergo all testing procedures.
* Able to read, understand, and complete study-related questionnaires
* Able to read and understand, and willing to sign the informed consent form (ICF).

Exclusion Criteria:

* Failure to provide informed consent.
* Any activity of daily living (ADL) disability (difficulty feeding, dressing, continence, bathing, toileting, and transferring).
* Lives in a nursing home; persons living in assisted or independent housing will not be excluded.
* Cognitive impairment, defined as a known diagnosis of dementia or Modified Mini-Mental State exam score <24
* Known neuromuscular or neurological conditions affecting somatosensory or motor function or control (e.g., hemiplegia, multiple sclerosis, peripheral neuropathy, Parkinson's disease, Myasthenia Gravis, Ataxia, Apraxia, post-polio syndrome, mitochondrial myopathy, etc.).
* Unable to communicate because of severe hearing loss or speech disorder.
* Severe visual impairment, which would preclude completion of the assessments.
* Cancer requiring treatment currently or in the past 2 years (except primary non-melanoma skin cancer or in situ cervical cancer)
* Hospitalization (medical confinement for ≥24 hours), or immobilization, or major surgical procedure requiring general anesthesia within 12 weeks prior to screening, or any planned surgical procedures during the study period.
* Chronic or relapsing/remitting gastrointestinal disorders such as inflammatory bowel disease and irritable bowel syndrome.
* Known history of human immunodeficiency virus (HIV) antibody at screening.
* Use of systemic glucocorticoids.
* Severe pulmonary disease, requiring either steroid pills or injections or the use of supplemental oxygen.
* Severe cardiac disease, including New York Heart Association (NYHA) Class III or IV congestive heart failure, clinically significant aortic stenosis, recent history of cardiac arrest (within 6-months), use of a cardiac defibrillator, or uncontrolled angina.
* Renal failure on hemodialysis
* Psychiatric conditions that warrant acute or chronic therapeutic intervention (e.g., major depressive disorder, bipolar disorder, panic disorder, schizophrenia) that in the investigators opinion may interfere with the conduct of study procedures
* Unable to undergo MRI or transcranial magnetic stimulation (TMS) (e. g. body containing any metallic medical devices or equipment, including heart pacemakers, metal prostheses, implants or surgical clips, any prior injury from shrapnel or grinding metal, exposure to metallic dusts, metallic shavings or having tattoos containing metallic dyes).
* Unable to reliably undergo exercise or strength tests described for this study.
* Participation in progressive resistance exercise within the previous 24 weeks prior to screening (for sub-studies only).
* Participation in any clinical trial within 12 weeks prior to screening (for sub-studies only).
* Limb amputation (except for toes) and/or any fracture within 24 weeks.
* Osteoarthritis, rheumatologic diseases or orthopedic disorders that will not allow completion of the motions required for the resistance exercise (for Resistance Exercise Training Sub-Study only).
* Conditions (such as myasthenia gravis, myositis, muscular dystrophy or myopathy, including drug-induced myopathy) leading to muscle loss, muscle weakness, muscle cramps or myalgia.
* Acute viral or bacterial upper or lower respiratory infection at screening
* Abnormal or uncontrolled blood pressure at the screening visit defined as diastolic BP >100 and/or systolic BP >170 mm Hg; if taking anti-hypertensive medication, have to be on stable doses of medication for more than 3 months.
* Medications known to alter the investigators' primary TMS-based outcomes. For instance, individuals taking benzodiazepines will be excluded from study participation.
* Current or recent history (within 1 year of screen) of heavy alcohol consumption or drug abuse that in the investigators opinion may interfere with the conduct of study procedures.
* Subjects with the following abnormal ECG findings at screening will be excluded: Electrocardiogram findings indicative of left ventricular hypertrophy (LVH) (based on Cornell voltage criteria):

  * For men: S in V3 plus R in a VL >2.8 milliVolts (mV) (28 mm)
  * For women: S in V3 plus R in a VL >2.0 mV (20 mm)
  * Electrocardiogram finding of QT prolongation

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2015-07; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Motor cortical excitability | Change from baseline measure after 12-weeks for resistance exercise group and 6-weeks for mental imagery and control groups.
  Obtained using transcranial magnetic stimulation
Voluntary activation | Change from baseline measure after 12-weeks for resistance exercise group and 6-weeks for mental imagery and control groups.
  Obtained based an the ratio of voluntary to electrically stimulated muscle forces

SECONDARY OUTCOMES:
White matter hyper intensities | Change from baseline measure after 12-weeks for resistance exercise group and 6-weeks for mental imagery and control groups.
  Obtained from brain MRI's
Stair climb power | Change from baseline measure after 12-weeks for resistance exercise group and 6-weeks for mental imagery and control groups.
  Time to ascend a flight of stairs
Motor unit discharge characteristics | Change from baseline measure after 12-weeks for resistance exercise group and 6-weeks for mental imagery and control groups.
  Obtained using decomposition EMG
Memory | Change from baseline measure after 12-weeks for resistance exercise group and 6-weeks for mental imagery and control groups.
  Memory assessed via the Repeatable Battery for the Assessment of Neuropsychological Status
Motor jerkiness | Change from baseline measure after 12-weeks for resistance exercise group and 6-weeks for mental imagery and control groups.
  Amount of variability in movement acceleration

CONTACTS AND LOCATIONS:
Overall Officials: Brian C Clark, PhD, Principal Investigator — Ohio University
Locations (1):
- Ohio Musculoskeletal and Neurological Institute (OMNI) at Ohio University, Athens, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tavoian D, Clark BC, Clark LA, Wages NP, Russ DW. Comparison of strategies for assessment of rate of torque development in older and younger adults. Eur J Appl Physiol. 2024 Feb;124(2):551-560. doi: 10.1007/s00421-023-05299-w. Epub 2023 Aug 25. PMID 37624389
- [Derived] Wages NP, Simon JE, Clark LA, Amano S, Russ DW, Manini TM, Clark BC. Relative contribution of muscle strength, lean mass, and lower extremity motor function in explaining between-person variance in mobility in older adults. BMC Geriatr. 2020 Jul 28;20(1):255. doi: 10.1186/s12877-020-01656-y. PMID 32723298
- See also: Ohio Musculoskeletal and Neurological Institute (OMNI) Website — http://www.ohio.edu/omni